CLINICAL TRIAL: NCT01178853
Title: Drug-Drug Interaction Study to Assess the Effects of Steady State Pitavastatin 4 mg or Rosuvastatin 40 mg on Steady-State Warfarin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NK-104-4.03US
Record Dates: First submitted 2010-08-09; First posted 2010-08-10 (Estimated); Results first posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Warfarin; Rosuvastatin Calcium; pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pitavastatin/Rosuvastatin (Experimental)
  Interventions: Drug: Warfarin; Drug: Warfarin 5mg + Rosuvastatin 40 mg once daily (QD); Drug: Warfarin 5 mg + Pitavastatin 4mg once daily (QD)
- Rosuvastatin/Pitavastatin (Experimental)
  Interventions: Drug: Warfarin; Drug: Warfarin 5mg + Rosuvastatin 40 mg once daily (QD); Drug: Warfarin 5 mg + Pitavastatin 4mg once daily (QD)

INTERVENTIONS:
Drug: Warfarin — Warfarin 5 mg once daily
Drug: Warfarin 5mg + Rosuvastatin 40 mg once daily (QD) — Warfarin 5mg + Rosuvastatin 40 mg once daily (QD)
Drug: Warfarin 5 mg + Pitavastatin 4mg once daily (QD) — Warfarin 5 mg + Pitavastatin 4mg

SUMMARY:
This is a Phase 4, single center, open label, 4 period, 2 treatment, crossover, drug-drug interaction study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy adult male or female volunteer aged 18 to 45 years, inclusive
* Subject has a body mass index of 18 to 32 kg/m2, inclusive
* Subject is able and willing to abstain from alcohol, grapefruit, caffeine
* Subject has no clinically relevant abnormalities on the basis of medical history, physical examination, and vital signs

Exclusion Criteria:

* Subject has clinically relevant out-of-range prothrombin time (PT), activated partial thromboplastin time, fibrinogen, protein C, or protein S
* Subject has abnormal prolongation of bleeding time at Screening
* Subject has hematuria on urinalysis
* Subject has personal or family history of coagulation or bleeding disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 July 2010 - 09 November 2010
Period: Period 1 (Warfarin Titration)
Arm/Group | Pitavastatin/Rosuvastatin | Rosuvastatin/Pitavastatin
Started | 24 | 24
Completed | 23 | 22
Not Completed | 1 | 2
Not completed — INR Out of Range | 1 | 2
Period: Period 2 (Warfarin + Study Drug)
Arm/Group | Pitavastatin/Rosuvastatin | Rosuvastatin/Pitavastatin
Started | 23 | 22
Completed | 22 | 22
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 3 (Warfarin Titration)
Arm/Group | Pitavastatin/Rosuvastatin | Rosuvastatin/Pitavastatin
Started | 22 | 22
Completed | 21 | 22
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 4 (Warfarin + Study Drug)
Arm/Group | Pitavastatin/Rosuvastatin | Rosuvastatin/Pitavastatin
Started | 21 | 22
Completed | 21 | 19
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin/Rosuvastatin | Rosuvastatin/Pitavastatin | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 24 | 48
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.4 (7.8) | 34.1 (7.2) | 33.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percent Mean Change From Baseline of International Normalized Ratio (INR)
Description: INR is the ratio of a patient's prothrombin time to a standard, raised to the power of the ISI value for the tissue factor reagent used (INR = (PT-Test/PT-Normal)^ISI)
Time Frame: 22 Days
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Warfarin + Pitavastatin | Warfarin + Rosuvastatin
Number analyzed (Participants) | 42 | 43
percent change | 0.0452 (2.61) | 0.1605 (9.43)

ADVERSE EVENTS:
Arm/Group | Warfarin + Pitavastatin | Warfarin + Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 6/42 | 3/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Warfarin + Pitavastatin (N=42) | Warfarin + Rosuvastatin (N=43)
Nausea (Gastrointestinal disorders) | 3 | 3
Headache (Nervous system disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
May not publish